CLINICAL TRIAL: NCT07235787
Title: Efficacy of Ultrasound Guided Microwave Ablation in the Treatment of Uterine Fibroids.
Acronym: MWAUF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jihad Hussien Mohamed Mahmoud (Other)
Responsible Party: Sponsor-Investigator, Jihad Hussien Mohamed Mahmoud, Specialist, Assiut University
Organization: Assiut University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ultrasound in uterine fibroids
Record Dates: First submitted 2025-11-16; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Uterine Fibroids (Leiomyoma); Symptomatic Uterine Leiomyoma
Keywords: Uterine fibroids; Leiomyoma; Microwave ablation (MWA); Ultrasound-guided ablation
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Intervention Model Description: This is described as a "prospective case series study" with all participants receiving the same intervention (microwave ablation).
Masking Description: This is an unmasked study. All participants and investigators know the intervention being performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Microwave Ablation Treatment (Experimental): Patients with symptomatic uterine fibroids who meet inclusion criteria will undergo ultrasound-guided percutaneous microwave thermal ablation (PMTA). The procedure involves percutaneous insertion of a microwave needle (1.4 to 1.6mm diameter and 15 to 20 cm length) into the fibroid under US guidance, with thermal ablation continuing for 10 to 30 minutes under IV sedation. Patients will be followed at 3 and 6 months to assess fibroid size reduction and symptom improvement.
  Interventions: Procedure: Ultrasound-Guided Percutaneous Microwave Thermal Ablation

INTERVENTIONS:
Procedure: Ultrasound-Guided Percutaneous Microwave Thermal Ablation — Minimally invasive percutaneous microwave thermal ablation of symptomatic uterine fibroids performed under ultrasound guidance. After 8 hours fasting and under aseptic conditions with IV sedation, a microwave needle (1.4-1.6mm diameter, 15-20cm length depending on fibroid site and size) is inserted percutaneously into the fibroid under ultrasound guidance. Thermal ablation is performed for 10-30 minutes to achieve coagulation necrosis of the fibroid tissue. Patients are discharged after several hours with post-procedure antibiotics and analgesics. Follow-up assessments at 3 and 6 months include ultrasound imaging, hemoglobin levels, and symptom evaluation.
  Other Names: PMTA; Microwave Ablation; MWA

SUMMARY:
Uterine fibroids are the most common benign tumors of the female genital tract and can significantly affect the quality of life in reproductive-age women, causing symptoms such as heavy menstrual bleeding, pelvic pressure, urinary disturbances, dyspareunia, and infertility. Traditional surgical interventions such as myomectomy and hysterectomy remain the standard of care, yet they are associated with considerable trauma, longer recovery times, and the loss of uterine function.

Microwave ablation (MWA) is a minimally invasive image-guided technique that uses microwave energy to induce coagulative necrosis in fibroid tissue, reducing its size and alleviating symptoms while preserving the uterus. This study aims to evaluate the feasibility, safety, and therapeutic effectiveness of ultrasound-guided percutaneous microwave thermal ablation (PMTA) in the management of symptomatic uterine fibroids.

Eligible participants are premenopausal women aged 25 years or older with symptomatic fibroids less than 10 cm in size and fewer than five in number. Exclusion criteria include pregnancy, bleeding disorders, chronic diseases contraindicating anesthesia, and ongoing anticoagulant therapy.

Each participant will undergo ultrasound-guided microwave ablation under aseptic conditions and sedation. Fibroid size, menstrual bleeding patterns, hemoglobin levels, and pain scores will be evaluated at baseline and during follow-up at 3 and 6 months. The primary outcome is the reduction in fibroid size, while secondary outcomes include symptom improvement and hemoglobin level changes.

This prospective case series will be conducted at Assiut University Hospitals, Egypt, with 20 participants referred from the Gynecology Department to the Interventional Radiology Unit. The results will provide valuable data on the clinical value of MWA as a uterus-preserving alternative for symptomatic uterine fibroids.

DETAILED DESCRIPTION:
This prospective interventional study will investigate the efficacy and safety of ultrasound-guided microwave ablation (MWA) for the treatment of uterine fibroids in premenopausal women who wish to avoid hysterectomy.

Fibroids are a leading cause of gynecologic morbidity and the most common indication for hysterectomy worldwide. Although medical and surgical therapies exist, many patients experience suboptimal outcomes or prefer minimally invasive, uterus-sparing treatments. MWA offers a promising alternative, providing precise thermal destruction of fibroid tissue through localized energy deposition with minimal collateral damage.

In this study, 20 women diagnosed with symptomatic uterine fibroids meeting inclusion criteria will be recruited. After pre-procedural evaluation-including clinical assessment, imaging, and laboratory testing-patients will undergo percutaneous MWA under ultrasound guidance. A microwave needle (1.4-1.6 mm in diameter and 15-20 cm in length) will be inserted into the fibroid, and thermal ablation will be applied for 10-30 minutes depending on lesion characteristics.

Post-procedure monitoring will include ultrasound assessment for immediate complications, with follow-up visits at 3 and 6 months to evaluate changes in fibroid size, menstrual characteristics, pain, and hemoglobin levels.

Statistical analysis will include descriptive measures and comparative tests (chi-square, t-test, or Wilcoxon rank-sum). Significance will be set at p ≤ 0.05. Data will be analyzed using STATA 13.

The study is conducted in compliance with the Declaration of Helsinki and has received ethical approval from the Assiut University Faculty of Medicine Ethics Committee. Written informed consent will be obtained from all participants prior to inclusion.

The expected outcome is to demonstrate that ultrasound-guided MWA is a feasible, safe, and effective minimally invasive therapy for uterine fibroids, potentially improving patient quality of life while avoiding the morbidity associated with hysterectomy and other surgical interventions.

ELIGIBILITY:
Inclusion Criteria:

Female patients aged 25 years or older Good general health Symptomatic uterine fibroids suitable for microwave ablation as determined by examining gynecologist Premenopausal status Acceptable risks for general anesthesia or sedation Number of fibroids: fewer than 5 Size of fibroid: less than 10 cm

Exclusion Criteria:

Ongoing anticoagulant treatment and/or known bleeding disorder Chronic diseases contraindicating general anesthesia Pregnancy Postmenopausal status 5 or more fibroids Fibroid size 10 cm or larger Poor general health precluding anesthesia or sedation

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Uterine Fibroid Size | Baseline, 3 months, and 6 months post-intervention
  Assessment of uterine fibroid dimensions (volume/diameter) measured by ultrasound imaging to evaluate the effectiveness of microwave ablation in reducing fibroid size.

SECONDARY OUTCOMES:
Change in Menstrual Bleeding | Baseline, 3 months, and 6 months post-intervention
  Assessment of menstrual bleeding severity measured by the number of pads/diapers used during menses and the number of days of menstruation.
Change in Hemoglobin Level | Baseline and 6 months post-intervention
  Assessment of hemoglobin (Hb) level through complete blood count (CBC) to evaluate improvement in anemia related to fibroid-associated bleeding.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Assiut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ierardi AM, Savasi V, Angileri SA, Petrillo M, Sbaraini S, Pinto A, Hanozet F, Marconi AM, Carrafiello G. Percutaneous High Frequency Microwave Ablation of Uterine Fibroids: Systematic Review. Biomed Res Int. 2018 Jan 8;2018:2360107. doi: 10.1155/2018/2360107. eCollection 2018. PMID 29511672
- [Result] Xia J, Teng D, Sui G, Luo Q, Lin Y, Wang H. Effectiveness and Safety of Ultrasound-guided Percutaneous Microwave Ablation for a Single Uterine Fibroid Greater than 300 cm3. J Minim Invasive Gynecol. 2023 Apr;30(4):290-299. doi: 10.1016/j.jmig.2022.12.013. Epub 2022 Dec 20. PMID 36563871